CLINICAL TRIAL: NCT06413667
Title: Assessment of the Alignment of the Atlas and Surrounding Tissues in Chronic Whiplash Associated Disorder
Acronym: MRAtlas
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Aart Nederveen, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2023.0628
Record Dates: First submitted 2024-04-15; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Chronic Whiplash Associated Disorder
Keywords: Atlas; MRI

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control participants: Healthy control participants without intervention
- Chronic Whiplash Associated Disorder: Chronic Whiplash Associated Disorder without intervention
- Tension headache: Tension headache without intervention

SUMMARY:
Whiplash is an injury caused by the rapid forward and backward movement of the neck, leading to injuries in bones or soft tissues, along with various symptoms. Recent studies indicate that muscles affected by whiplash may show increased fat buildup and reduced muscle volume. However, these changes in muscle do not completely account for the pain and other symptoms reported. Besides soft tissues, whiplash can also injure bone structures, including the cervical spine. Until now, studies focused mainly on fractures of the cervical spine, often overlooking the position and alignment of the atlas and dens (C1 and C2). The aim of this study is to evaluate the position and alignment of the Atlas in chronic whiplash-associated disorder (grades 1 or 2) and compare it to patients with tension headache and healthy controls. Additionally, it will explore how these factors relate to pain intensity, neck movement limitations, daily activities, overall improvement, and quality of life.

DETAILED DESCRIPTION:
Treating some neurological conditions, like chronic whiplash-associated disorder (WAD), is highly challenging for medical practitioners. Patients with chronic WAD frequently visit their general practitioner because it's hard to pinpoint the cause of their symptoms. This makes finding the right treatment very difficult. The number of chronic WAD cases is rising worldwide, costing Europe an estimated 10 billion euros annually. Half of all whiplash injuries develop into chronic conditions, leading to significant disability and societal costs. These patients face major limitations in daily activities, greatly affecting their quality of life.

Whiplash is an injury caused by the rapid forward and backward movement of the neck, leading to injuries in bones or soft tissues, along with various symptoms. Recent studies indicate that muscles affected by whiplash may show increased fat buildup and reduced muscle volume. However, these changes in muscle do not completely account for the pain and other symptoms reported. Besides soft tissues, whiplash can also injure bone structures, including the cervical spine. Until now, studies focused mainly on fractures of the cervical spine, often overlooking the position and alignment of the atlas and dens (C1 and C2).

The aim of this study is to apply advanced imaging technologies to assess the position and alignment of the Atlas (C1) and the surrounding tissues. The study has three main goals:

i. Study the feasibility and repeatability of state-of-the-art MRI measurements in 30 healthy controls across an age range of 18 to 75 years.

ii. Assess the position and alignment of the Atlas and surrounding tissues using MRI in patients with WAD, compared to patients with tension headaches and healthy control participants;

iii. Relate these MRI parameters to neurological examinations and questionnaires (patient- reported outcome measures) in patients with WAD and tension headaches.

ELIGIBILITY:
Inclusion Criteria: Participants fulfilling the criteria mentioned below:

Control participants In order to be eligible to participate in this study, a participant must meet the following criteria:

* Healthy individuals
* Ability to follow test instructions
* Aged between 18 - 75 years

Chronic Whiplash Associated Disorder

In order to be eligible to participate in this study, a participant must meet the following criteria:

* Healthy individuals
* Ability to follow test instructions
* WAD 1 or 2 Diagnosis
* Aged between 18 - 75 years

Tension headache

In order to be eligible to participate in this study, a participant must meet the following criteria:

* Healthy individuals
* Ability to follow test instructions
* Diagnosis Tension headache
* Aged between 18 -75 years

Exclusion Criteria: A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Inability to provide informed consent
* Have a history of claustrophobia
* Patient/ participant is not eligible to follow instructions
* Contra-indication for MRI (e.g., pacemaker, claustrophobia)
* Being under investigation for non-diagnosed disease at the time of investigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to evaluate high resolution MR techniques to measure position and alignment of the Atlas and its surrounding structures in healthy participants, individuals with tension headache and individuals with chronic whiplash disorder.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Repeatability measurement | 12 months
  MRI images will be used to measure the angles between the Atlas and adjacent vertebrae at two different time points in the same healthy participants.
Alignment of the Atlas | 12 months
  MRI images will be used to measure the angles between the Atlas and adjacent vertebrae in the patient groups.
Neurological examination scores | 18 months
  A neurological examination will be performed and scored during the participants' visit
Quality of life scores | 18 months
  The scores will be obtained by using quality of life questionnaire

SECONDARY OUTCOMES:
Muscle volume | 24 months
  Muscle volume (in mm3) will be measured from the quantitative MRI scans and compared across the groups.
Fat fraction | 24 months
  Fat fraction (in %) will be measured from MRI and compared across the groups.
Blood flow | 24 months
  Blood flow (in cm/s) in the brain feeding arteries will be obtained from the quantitative MRI scans and compared across the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands